CLINICAL TRIAL: NCT01208103
Title: Phase II Study of Bevacizumab Combined With Capecitabine and Oxaliplatin (CAPOX) in Patients With Advanced Adenocarcinoma of the Small Bowel or Ampulla of Vater
Brief Title: Bevacizumab, Capecitabine, and Oxaliplatin in Treating Advanced Small Intestinal or Ampulla of Vater Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0626; NCI-2018-01828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2011-00470; 2009-0626 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2010-08-31; First posted 2010-09-23 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Ampulla of Vater Adenocarcinoma; Small Intestinal Adenocarcinoma; Stage III Ampulla of Vater Cancer AJCC v8; Stage III Small Intestinal Adenocarcinoma AJCC v8; Stage IIIA Ampulla of Vater Cancer AJCC v8; Stage IIIA Small Intestinal Adenocarcinoma AJCC v8; Stage IIIB Ampulla of Vater Cancer AJCC v8; Stage IIIB Small Intestinal Adenocarcinoma AJCC v8; Stage IV Ampulla of Vater Cancer AJCC v8; Stage IV Small Intestinal Adenocarcinoma AJCC v8
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (oxaliplatin, bevacizumab, capecitabine) (Experimental): Participants receive oxaliplatin via CVC over 2 hours and bevacizumab IV over 30-90 minutes on day 1. Participants also receive capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Oxaliplatin — Given CVC
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669

SUMMARY:
This phase II trial studies how well bevacizumab given with capecitabine and oxaliplatin work in treating participants with small bowel or ampulla of Vater adenocarcinoma that has spread to other places in the body. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Drugs using in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving bevacizumab, capecitabine, and oxaliplatin may work better in treating participants with small intestinal or ampulla of Vater adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival (PFS) at six months for patients with advanced adenocarcinoma of the small bowel (small intestine) or ampulla of Vater treated with capecitabine, oxaliplatin (CAPOX) and bevacizumab.

SECONDARY OBJECTIVES:

I. To determine the response rate (RR) for CAPOX and bevacizumab. II. To determine the overall progression free survival for CAPOX and bevacizumab.

III. To determine the overall survival (OS) for CAPOX and bevacizumab. IV. To determine the toxicity of CAPOX and bevacizumab.

OUTLINE:

Participants receive oxaliplatin via central venous catheter (CVC) over 2 hours and bevacizumab intravenously (IV) over 30-90 minutes on day 1. Participants also receive capecitabine orally (PO) twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 10 and 30 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the small bowel or ampulla of Vater
* Prior adjuvant chemotherapy (including fluorouracil [5-FU], capecitabine, and oxaliplatin) for the treatment of adenocarcinoma of the small bowel or ampulla of Vater is allowed if completed >= 52 weeks prior to first dose of study treatment
* Prior capecitabine or 5-FU administered as a radio-sensitizing agent concurrently with external beam radiotherapy is allowed
* Patients must have metastatic disease
* A minimum of 4 weeks must have elapsed from completion of any prior chemotherapy or radiotherapy or surgery and the start date of study therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * In patients with known Gilbert's syndrome direct bilirubin =< 1.5 x ULN will be used as organ function criteria, instead of total bilirubin
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 x ULN
* Calculated creatinine clearance (CrCl) > 50 cc/min (calculated using the Cockcroft and Gault formula)
* Negative serum or urine pregnancy test in women with childbearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization), within one week prior to initiation of treatment
* Patients must sign an Informed Consent and Authorization indicating that they are aware of the investigational nature of this study and the known risks involved
* The effects of the combination of CAPOX and bevacizumab on the developing fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and for six months following the completion of therapy. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with oxaliplatin or capecitabine or bevacizumab, breast feeding must be discontinued

Exclusion Criteria:

* Patients who have received prior chemotherapy for their metastatic disease are excluded. Chemotherapy if given as a radiation-sensitizer is allowed
* Patients may not be receiving any other investigational agents nor have received any investigational drug 28 days prior to enrollment
* Known history of dihydropyrimidine (DPD) deficiency
* Peripheral neuropathy of grade 3 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* Because of the interaction between coumadin and capecitabine, patients taking therapeutic doses of coumadin-derivative anticoagulants are not eligible. Low-dose coumadin (e.g. 1 mg PO per day) in patients with in-dwelling venous access devices is allowed but increased frequency of international normalized ratio (INR) monitoring is recommended
* Prior treatment with bevacizumab or known hypersensitivity to any component of bevacizumab
* Inadequately controlled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* New York Heart Association (NYHA) grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to day 1
* History of stroke or transient ischemic attack within 6 months prior to day 1.
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1
* History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month prior to day 1
* History of abdominal fistula or gastrointestinal perforation which must have resolved at least 6 months prior to day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure excluding placement of a vascular access device, within 7 days prior to day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening as demonstrated by either (1) urine protein:creatinine (UPC) ratio of >= 1.0 or (2) urine dipstick for proteinuria >= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis should undergo a 24 hour urine collection and must demonstrate =< 1g of protein in 24 hours to be eligible)
* Known central nervous system (CNS) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; gamma knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician
* Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than this study
* Pregnancy (positive pregnancy test) or lactation
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix, within last five years
* Inability to comply with study and/or follow-up procedures
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05-06 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2011 to November 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Bevacizumab + Capecitabine + Oxaliplatin: Capecitabine 750 mg/m2 oral twice daily, Days 1 - 14 and Bevacizumab 7.5 mg/kg IV over 90 minutes on Day 1 and Oxaliplatin 130 mg/m2 IV over 2 hours Day 1 of 21-day cycle.
Period: Overall Study
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Started | 30
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival (PFS) at Six Months
Description: A Bayesian sequential monitoring design will be used. PFS will be estimated using the Kaplan-Meier method.The length of time interval in months from date of first treatment, during and after the treatment a participant lives without progression.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bevacizumab + Capecitabine + Oxaliplatin: Capecitabine 750mg/m2 oral twice daily, Days 1 - 14 and Panitumumab 9 mg/kg IV over 60 minutes on Day 1 and Oxaliplatin 130 mg/m2 IV over 2 hours Day 1 of 21-day cycle.
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Number analyzed (Participants) | 30
percentage of participants | 68 [52 to 88]

2. Secondary Outcome: To Determine the Response Rate (RR) for CAPOX and Bevacizumab
Description: Complete response + Partial response using RECIST 1.1 (Response Evaluation Criteria in Solid Tumor)
Time Frame: 39 months
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab + Capecitabine + Oxaliplatin: Capecitabine 750mg/m2 oral twice daily, Days 1 - 14 and Bevacizumab 7.5 mg/kg IV over 90 minutes on Day 1 and Oxaliplatin 130 mg/m2 IV over 2 hours Day 1 of 21-day cycle.
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Number analyzed (Participants) | 30
Participants
  Complete Response | 1
  Partial Response | 13
  Stable Disease | 10
  Progressive Disease | 5
  Unevaluable | 1

3. Secondary Outcome: To Determine the Overall PFS for CAPOX and Bevacizumab
Description: Time interval in months from date of first treatment until the date of first documented progression
Time Frame: 39 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Number analyzed (Participants) | 30
months | 8.7 [4.9 to 10.5]

4. Secondary Outcome: To Determine the Overall Survival (OS) for CAPOX and Bevacizumab
Description: The length of time interval in months from date of first treatment until the date of death or lost follow-up
Time Frame: 39 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Number analyzed (Participants) | 30
months | 12.9 [9.2 to 19.7]

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicity was graded according to the NCI Common terminology Criteria for Adverse Events (CTCAE) 4.0 except for neurosensory and skin toxicity. Neurosensory toxicity was graded according to the Neurologic Toxicity Scale for Oxaliplatin Dose Adjustments.
Time Frame: 39 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
Number analyzed (Participants) | 30
participants | 30

ADVERSE EVENTS:
Time Frame: Assessed up to 67 months
Arm/Group | Bevacizumab + Capecitabine + Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 30/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Capecitabine + Oxaliplatin (N=30)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Capecitabine + Oxaliplatin (N=30)
Anemia (Blood and lymphatic system disorders) | 17
Platelet count decreased (Investigations) | 14
Neutrophil count decreased (Investigations) | 11
Abdominal pain (Gastrointestinal disorders) | 7
Alanine aminotransferase increased (Investigations) | 16
Alkaline phosphatase increased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 23
Ascites (Gastrointestinal disorders) | 1
Aspartate (Investigations) | 21
Blood bilirubin increased (Investigations) | 6
Colitis (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 11
Diarrhea (Gastrointestinal disorders) | 23
Dysesthesia (Nervous system disorders) | 26
Fatigue (General disorders) | 24
Headache (Nervous system disorders) | 3
Hypertension (Vascular disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 3
Nausea (Gastrointestinal disorders) | 23
Pancreatitis (Gastrointestinal disorders) | 1
Peripheral sensor neuropathy (Nervous system disorders) | 23
Pnuemonitis (Respiratory, thoracic and mediastinal disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Proteinuria (Renal and urinary disorders) | 12
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Weight loss (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT01208103/Prot_SAP_000.pdf